CLINICAL TRIAL: NCT04366349
Title: A Randomized, Double-blind, Single Ascending Dose Study to Determine the Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of GSK3772847 Administered Subcutaneously in Healthy Participants
Brief Title: A Study to Evaluate the Safety and Tolerability, Pharmacokinetics (PK) and Pharmacodynamics (PD) of Melrilimab (GSK3772847) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 209635
Record Dates: First submitted 2020-04-27; First posted 2020-04-28 (Actual); Results first posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-09

CONDITIONS: Healthy Volunteers; Asthma
Keywords: Pharmacokinetics; Pharmacodynamics; Safety; GSK3772847; Tolerability
MeSH Terms: conditions — Asthma | interventions — melrilimab

STUDY DESIGN:
Intervention Model Description: This is a single arm study.
Who Masked: Participant, Investigator
Masking Description: This is a double blind study and participants and investigator will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Participants receiving melrilimab (GSK3772847) 70 milligram (mg) (Experimental): Participants will receive a single dose of melrilimab (GSK3772847) 70 milligram (mg) subcutaneously (SC) injection by an health care professional (HCP).
  Interventions: Biological: melrilimab (GSK3772847) 70 milligram (mg)
- Participants receiving melrilimab (GSK3772847) 140 milligram (mg) (Experimental): Participants will receive a single dose of melrilimab (GSK3772847) 140 milligram (mg) subcutaneously (SC) injection by an health care professional (HCP).
  Interventions: Biological: melrilimab (GSK3772847) 140 milligram (mg)
- Participants receiving Placebo (Placebo Comparator): Participants will receive a single dose of placebo subcutaneously (SC) injection by an health care professional (HCP).
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: melrilimab (GSK3772847) 70 milligram (mg) — melrilimab (GSK3772837) will be available at a dose strength of 70 milligram per milliliter (mg/mL) in a 3 milliliter (mL) glass vial.
  Arms: Participants receiving melrilimab (GSK3772847) 70 milligram (mg)
Biological: melrilimab (GSK3772847) 140 milligram (mg) — Two doses of melrilimab (GSK3772837) 70 milligram per milliliter (mg/mL) will be administered to achieve a dose strength of 140 milligram per milliliter (mg/mL)
  Arms: Participants receiving melrilimab (GSK3772847) 140 milligram (mg)
Other: Placebo — Placebo to match melrilimab (GSK3772847) will be available in the form of solution for injection in a 3 milliliter (mL) glass vial.
  Arms: Participants receiving Placebo

SUMMARY:
GSK3772847, an anti-interleukin (IL) 33-receptor monoclonal antibody, is a novel treatment for asthma. The purpose of this study to evaluate the safety and tolerability, PK and PD of single ascending doses of GSK3772847 administered subcutaneously (SC) to healthy participants. This study will also establish the bioavailability of SC formulation and evaluate the safety in particular injection site tolerability of route. Participants will either receive a single dose of 70 milligram (mg) GSK3772847 or placebo in (Cohort 1) and 140 mg GSK3772847 or placebo in Cohorts 2, 3 (Japanese participants) and 4 (Chinese participants). The site of injection will be upper arm; abdomen or thigh for cohorts 1 and 2 with cohorts 3 and 4 will receive injections in the upper arm only. Approximately, the total duration of study will be up to 89 days.

ELIGIBILITY:
Inclusion Criteria:

* Participants age in between 18 to 65 years, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring. A participant with a clinical abnormality or laboratory parameters not specifically listed in the exclusion criteria that is outside the reference range for the population being studied may be included only if the investigator, in consultation with the Medical Monitor (if required), agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures or results.
* Japanese participants are eligible based on meeting all of the following criteria: healthy male and female participants born in Japan; are descendants of four ethnic Japanese grandparents and two ethnic Japanese parents; holding a Japanese passport or identity papers; being able to speak Japanese; have lived outside Japan for less than 10 years at the time of screening.
* Chinese Participants are eligible based on meeting all of the following: healthy male and female participants born in mainland China; are descendants of four Chinese grandparents and two Chinese parents; holding a Chinese passport or identity papers; being able to speak Chinese; have lived outside China for less than 10 years at the time of screening; Body weight 35-150 kilogram (kg) and body mass index (BMI) within the range 18-32 kilogram per square meter (kg/m2) (inclusive).
* Female participant: A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies; is not a woman of childbearing potential (WOCBP) or is a WOCBP and using an acceptable contraceptive method during the intervention period (at a minimum until after the last dose of study intervention); the investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention; a WOCBP must have a negative highly sensitive pregnancy test ([urine] as required by local regulations) within 24 hours before the first dose of study intervention; if a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required,. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive; additional requirements for pregnancy testing during and after study intervention are located; The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Alanine transaminase (ALT) >2 times of (x) upper limit of normal (ULN).
* Bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent [%]).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Ongoing or recurrent infections.
* QT interval corrected for heart rate by Fridericia's formula (QTcF) >450 millisecond (msec) or any of the following abnormal and clinically significant electrocardiogram (ECG) findings; sinus bradycardia <45 beats per minute (bpm); sinus tachycardia >=110 bpm; multifocal atrial tachycardia (wandering atrial pacemaker with rate >100 bpm); evidence of Mobitz II second degree or third degree atrioventricular (AV) block; pathological Q waves (defined as wide [>0.04 seconds] and deep [>0.4 millivolt (mV) (4 millimeter (mm) with 10mm/mV setting)] or >25% of the height of the corresponding R wave, providing the R wave was >0.5 mV [5 mm with 10mm/mV setting], appearing in at least two contiguous leads; Evidence of ventricular ectopic couplets, bigeminy, trigeminy or multifocal premature ventricular complexes; For participants without complete right bundle branch block: QT interval corrected for heart rate by Fridericia's formula (QTc[F]) >=450 msec or an ECG that is unsuitable for QT measurements (e.g., poor defined termination of the T wave); for participants with complete right bundle branch block: QTc(F) >=480 msec or an ECG that is unsuitable for QT measurements (e.g., poor defined termination of the T wave); ST-T wave abnormalities (excluding non-specific ST-T wave abnormalities); Clinically significant conduction abnormalities (e.g., Wolff-Parkinson-White syndrome or bifascicular block defined as complete left bundle branch block or complete right bundle branch block with concomitant left fascicular block); Clinically significant arrhythmias (e.g., atrial fibrillation with rapid ventricular response, ventricular tachycardia).
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including saint [St] John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) before the first dose of study medication and until study completion, unless in the opinion of the investigator and GlaxoSmithKline (GSK) Medical Monitor the medication will not interfere with the study procedures or compromise participant safety.
* The participant has been in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Presence of Hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to first dose of study intervention.
* Positive Hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention.
* Positive Hepatitis C ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study intervention.
* A positive test for human immunodeficiency virus (HIV) antibody.
* Where participation in the study would result in donation of blood or blood products in excess of 500 milliliter (mL) within 3 months.
* A positive pre-study drug/alcohol screen.
* Any history of substance abuse or a positive test for drugs of abuse at screening or admission.
* Known, pre-existing parasitic infestations within 6 months prior to Screening.
* Vaccinated with live or attenuated vaccines within 4 weeks prior to receiving investigational product (IP) and up to 6 months after dose administration of GSK3772847.
* A positive highly sensitive pregnancy test (urine or serum as required by local regulations) at screening.
* Positive urinary cotinine test indicative of smoking history at screening or each in-house admission to the clinical research unit or regular use of tobacco- or nicotine-containing products (e.g. nicotine patches or vaporizing devices) within 6 months prior to screening.
* Participants with allergy or intolerance to a monoclonal antibody or biologic or to any components of the formulation used in this study.
* A vulnerable participant. defined as individuals whose willingness to volunteer in a clinical trial may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate.
* Participants who work for the Sponsor, contract research organization (CRO), or one of the study centers.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2020-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Pefani E, Stone S, Zhu CQ, Nunn C, Fairman D. Safety, tolerability, and pharmacokinetics of a single ascending subcutaneous dose of GSK3772847 in healthy participants. Pharmacol Res Perspect. 2023 Apr;11(2):e01054. doi: 10.1002/prp2.1054. PMID 36846967

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who met the eligibility criteria were assigned to one of the four cohorts and were randomly allocated within each cohort to receive a single dose of either GSK3772847 or placebo. All treatments were administered subcutaneously. The site of injection was randomized to the upper arm, abdomen, or thigh for cohorts 1 and 2. Injection was given in the upper arm only in cohorts 3 and 4.
Pre-assignment Details: A total of 65 participants were enrolled in this study.
Groups:
- Cohorts 1 and 2: Placebo SC: Participants received a single dose of placebo subcutaneous (SC) injection in the upper arm, abdomen or thigh by a health care professional in Cohorts 1 and 2.
- Cohort 1: GSK3772847 70 mg SC: Participants received a single dose of GSK3772847 70 milligram (mg) SC injection in the upper arm, abdomen or thigh by a health care professional in Cohort 1.
- Cohort 2: GSK3772847 140 mg SC: Participants received a single dose of GSK3772847 140 mg SC injection in the upper arm, abdomen or thigh by a health care professional in Cohort 2.
- Cohorts 3 and 4: Placebo SC: Japanese and Chinese participants received a single dose of placebo SC injection in the upper arm by a health care professional in Cohorts 3 and 4.
- Cohort 3: GSK3772847 140 mg SC in Japanese Participants: Japanese participants received a single dose of GSK3772847 140 mg SC injection in the upper arm by a health care professional in Cohort 3.
- Cohort 4: GSK3772847 140 mg SC in Chinese Participants: Chinese participants received a single dose of GSK3772847 140 mg SC injection in the upper arm by a health care professional in Cohort 4.
Period: Overall Study
Arm/Group | Cohorts 1 and 2: Placebo SC | Cohort 1: GSK3772847 70 mg SC | Cohort 2: GSK3772847 140 mg SC | Cohorts 3 and 4: Placebo SC | Cohort 3: GSK3772847 140 mg SC in Japanese Participants | Cohort 4: GSK3772847 140 mg SC in Chinese Participants
Started | 13 | 18 | 18 | 4 | 6 | 6
Completed | 12 | 18 | 18 | 4 | 6 | 6
Not Completed | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohorts 1 and 2: Placebo SC | Cohort 1: GSK3772847 70 mg SC | Cohort 2: GSK3772847 140 mg SC | Cohorts 3 and 4: Placebo SC | Cohort 3: GSK3772847 140 mg SC in Japanese Participants | Cohort 4: GSK3772847 140 mg SC in Chinese Participants | Total
Number analyzed (Participants) | 13 | 18 | 18 | 4 | 6 | 6 | 65
Age, Customized [Count of Participants; unit: Participants]
  18-64 years | 13 | 18 | 18 | 4 | 6 | 6 | 65
  >=65-84 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  >=85 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 9 | 4 | 5 | 1 | 33
  Male | 7 | 10 | 9 | 0 | 1 | 5 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 4 | 5 | 2 | 0 | 0 | 0 | 11
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White: White/Caucasian/European Heritage | 8 | 13 | 14 | 0 | 0 | 0 | 35
  Asian: Central/South Asian Heritage | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian: East Asian Heritage | 0 | 0 | 0 | 2 | 0 | 6 | 8
  Asian: Japanese Heritage | 0 | 0 | 0 | 2 | 6 | 0 | 8
  Asian: South East Asian Heritage | 0 | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A SAE is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, and other situations which involve medical or scientific judgment.
Time Frame: Up to Day 85
Population: Safety Population consisted of all randomized participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1 and 2: Placebo SC | Cohort 1: GSK3772847 70 mg SC | Cohort 2: GSK3772847 140 mg SC | Cohorts 3 and 4: Placebo SC | Cohort 3: GSK3772847 140 mg SC in Japanese Participants | Cohort 4: GSK3772847 140 mg SC in Chinese Participants
Number analyzed (Participants) | 13 | 18 | 18 | 4 | 6 | 6
Participants
  AEs | 3 | 2 | 3 | 1 | 2 | 2
  SAEs | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Area Under the Plasma Concentration Time Curve From 0 to t (AUC[0-t]) of GSK3772847
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3772847. Pharmacokinetic Population consisted of all randomized participants who received at least one dose of study treatment, and for whom at least one pharmacokinetic sample was obtained, analyzed and measurable.
Time Frame: Day 1: Pre-dose, 2, 4, 8 hours post-dose; Days 2, 3, 4, 5, 6, 9, 15, 29, 43, 57, 71 and 85
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cohort 1: GSK3772847 70 mg SC | Cohort 2: GSK3772847 140 mg SC | Cohort 3: GSK3772847 140 mg SC in Japanese Participants | Cohort 4: GSK3772847 140 mg SC in Chinese Participants
Number analyzed (Participants) | 18 | 18 | 6 | 6
Hours*microgram per milliliter | 4139.092 (34.1) | 10271.279 (25.2) | 13356.462 (29.7) | 11285.792 (25.4)

3. Primary Outcome: Area Under the Plasma Concentration Time Curve From Time Zero to Infinity (AUC[0-infinity]) of GSK3772847
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3772847.
Time Frame: Day 1: Pre-dose, 2, 4, 8 hours post-dose; Days 2, 3, 4, 5, 6, 9, 15, 29, 43, 57, 71 and 85
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*microgram per milliliter
Arm/Group | Cohort 1: GSK3772847 70 mg SC | Cohort 2: GSK3772847 140 mg SC | Cohort 3: GSK3772847 140 mg SC in Japanese Participants | Cohort 4: GSK3772847 140 mg SC in Chinese Participants
Number analyzed (Participants) | 18 | 18 | 6 | 6
Hours*microgram per milliliter | 4336.865 (32.9) | 10575.235 (25.2) | 13936.982 (34.0) | 11576.445 (26.6)

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of GSK3772847
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3772847.
Time Frame: Day 1: Pre-dose, 2, 4, 8 hours post-dose; Days 2, 3, 4, 5, 6, 9, 15, 29, 43, 57, 71 and 85
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Cohort 1: GSK3772847 70 mg SC | Cohort 2: GSK3772847 140 mg SC | Cohort 3: GSK3772847 140 mg SC in Japanese Participants | Cohort 4: GSK3772847 140 mg SC in Chinese Participants
Number analyzed (Participants) | 18 | 18 | 6 | 6
Microgram per milliliter | 7.8276 (38.4) | 15.0569 (24.5) | 15.9309 (25.5) | 15.8324 (15.2)

5. Primary Outcome: Time to Cmax (Tmax) of GSK3772847
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3772847.
Time Frame: Day 1: Pre-dose, 2, 4, 8 hours post-dose; Days 2, 3, 4, 5, 6, 9, 15, 29, 43, 57, 71 and 85
Population: Pharmacokinetic Population.
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: GSK3772847 70 mg SC | Cohort 2: GSK3772847 140 mg SC | Cohort 3: GSK3772847 140 mg SC in Japanese Participants | Cohort 4: GSK3772847 140 mg SC in Chinese Participants
Number analyzed (Participants) | 18 | 18 | 6 | 6
Hours | 120.000 [48.00 to 382.42] | 130.358 [71.95 to 311.80] | 146.175 [144.93 to 312.63] | 204.925 [72.00 to 381.65]

6. Primary Outcome: Apparent Terminal Half-life (t1/2) of GSK3772847
Description: Blood samples were collected at indicated time points for pharmacokinetic analysis of GSK3772847.
Time Frame: Day 1: Pre-dose, 2, 4, 8 hours post-dose; Days 2, 3, 4, 5, 6, 9, 15, 29, 43, 57, 71 and 85
Population: Pharmacokinetic Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | Cohort 1: GSK3772847 70 mg SC | Cohort 2: GSK3772847 140 mg SC | Cohort 3: GSK3772847 140 mg SC in Japanese Participants | Cohort 4: GSK3772847 140 mg SC in Chinese Participants
Number analyzed (Participants) | 18 | 18 | 6 | 6
Hours | 243.275 (17.1) | 293.144 (27.6) | 342.622 (36.8) | 291.690 (22.2)

7. Secondary Outcome: Maximal Decrease in Ratio to Baseline in Free Soluble Suppressor of Tumorigenicity 2 (ST2) Concentration
Description: Blood samples were collected to measure free soluble ST2 concentration. Maximal decrease from Baseline was the largest decrease calculated across all time points post dose. Ratio to Baseline is defined as post-dose visit value divided by Baseline value. Baseline was the most recent recorded value before dosing on Day 1 (Pre-dose). Pharmacodynamic Population consisted of all randomized participants who received at least one dose of study treatment, and for whom at least one pharmacokinetic sample was obtained, analyzed and measurable.
Time Frame: Baseline and up to Day 85/early withdrawal
Population: Pharmacodynamic Population. Only those participants with data available at indicated time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cohorts 1 and 2: Placebo SC | Cohort 1: GSK3772847 70 mg SC | Cohort 2: GSK3772847 140 mg SC | Cohorts 3 and 4: Placebo SC | Cohort 3: GSK3772847 140 mg SC in Japanese Participants | Cohort 4: GSK3772847 140 mg SC in Chinese Participants
Number analyzed (Participants) | 11 | 18 | 18 | 4 | 6 | 6
Ratio | 0.7573 [0.6586 to 0.9660] | 0.0621 [0.0512 to 0.0871] | 0.0417 [0.0372 to 0.0511] | 0.8073 [0.7150 to 0.9028] | 0.0453 [0.0311 to 0.0638] | 0.0433 [0.0399 to 0.0469]

8. Secondary Outcome: Maximal Increase in Ratio to Baseline in Total Soluble ST2 Concentration
Description: Blood samples were collected to measure total soluble ST2 concentration. Maximal increase from Baseline was the largest increase calculated across all timepoints post dose. Ratio to Baseline is defined as post-dose visit value divided by Baseline value. Baseline was the most recent recorded value before dosing on Day 1 (Pre-dose).
Time Frame: Baseline and up to Day 85/early withdrawal
Population: Pharmacodynamic Population. Only those participants with data available at indicated time points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cohorts 1 and 2: Placebo SC | Cohort 1: GSK3772847 70 mg SC | Cohort 2: GSK3772847 140 mg SC | Cohorts 3 and 4: Placebo SC | Cohort 3: GSK3772847 140 mg SC in Japanese Participants | Cohort 4: GSK3772847 140 mg SC in Chinese Participants
Number analyzed (Participants) | 12 | 18 | 18 | 4 | 6 | 6
Ratio | 2.0573 [-1.8417 to 10.8808] | 25.4604 [22.1566 to 31.4077] | 40.6790 [9.4889 to 112.2080] | 1.7203 [1.1951 to 2.2921] | 39.1039 [29.7883 to 50.6161] | 45.7791 [35.8528 to 57.6231]

9. Secondary Outcome: Number of Participants With Confirmed Positive Anti-GSK3772847 Antibodies
Description: Serum samples were collected at indicated time points and analyzed for the presence of anti-GSK3772847 antibodies using a tiered approach including a screening assay, a confirmation assay and calculation of titer.
Time Frame: Days 1, 15, 29, 57 and 85/early withdrawal
Population: Pharmacodynamic Population. Only those participants with data available at indicated time points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohorts 1 and 2: Placebo SC | Cohort 1: GSK3772847 70 mg SC | Cohort 2: GSK3772847 140 mg SC | Cohorts 3 and 4: Placebo SC | Cohort 3: GSK3772847 140 mg SC in Japanese Participants | Cohort 4: GSK3772847 140 mg SC in Chinese Participants
Number analyzed (Participants) | 13 | 18 | 18 | 4 | 6 | 6
Participants
  Day 1: n=13,18,18,4,6,6 | 0 | 0 | 0 | 0 | 0 | 0
  Day 15: n=13,18,18,4,6,6 | 0 | 0 | 0 | 0 | 0 | 0
  Day 29: n=12,18,17,4,6,6: number analyzed (Participants) | 12 | 18 | 17 | 4 | 6 | 6
  Day 29: n=12,18,17,4,6,6 | 0 | 0 | 0 | 0 | 0 | 0
  Day 57: n=12,18,18,4,6,6: number analyzed (Participants) | 12 | 18 | 18 | 4 | 6 | 6
  Day 57: n=12,18,18,4,6,6 | 0 | 0 | 0 | 0 | 0 | 1
  Day 85/early withdrawal: n=12,18,18,4,6,6: number analyzed (Participants) | 12 | 18 | 18 | 4 | 6 | 6
  Day 85/early withdrawal: n=12,18,18,4,6,6 | 0 | 0 | 0 | 0 | 0 | 1

10. Secondary Outcome: Ratio to Baseline in Plasma 4 Beta-hydroxy (4BetaOH) Cholesterol/Cholesterol
Description: Blood samples were collected at indicated time points to measure 4BetaOH cholesterol/cholesterol. Ratio to Baseline is defined as post-dose visit value divided by Baseline value. Baseline value was the latest pre-dose assessment (Day 1 Pre-dose).
Time Frame: Baseline, Days 5, 15, 29 and 85/early withdrawal
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Cohorts 1 and 2: Placebo SC | Cohort 1: GSK3772847 70 mg SC | Cohort 2: GSK3772847 140 mg SC | Cohorts 3 and 4: Placebo SC | Cohort 3: GSK3772847 140 mg SC in Japanese Participants | Cohort 4: GSK3772847 140 mg SC in Chinese Participants
Number analyzed (Participants) | 13 | 18 | 18 | 4 | 6 | 6
Ratio
  Day 5: n=13,18,18,4,6,6 | 1.117 [0.979 to 1.274] | 0.998 [0.945 to 1.053] | 1.092 [0.976 to 1.221] | 1.062 [0.580 to 1.944] | 1.051 [0.951 to 1.163] | 1.192 [0.941 to 1.511]
  Day 15: n=11,18,18,4,6,6: number analyzed (Participants) | 11 | 18 | 18 | 4 | 6 | 6
  Day 15: n=11,18,18,4,6,6 | 1.021 [0.883 to 1.180] | 0.992 [0.914 to 1.076] | 1.092 [0.958 to 1.244] | 1.106 [0.790 to 1.547] | 1.054 [0.892 to 1.244] | 1.285 [1.050 to 1.572]
  Day 29: n=12,18,17,4,6,6: number analyzed (Participants) | 12 | 18 | 17 | 4 | 6 | 6
  Day 29: n=12,18,17,4,6,6 | 1.119 [0.942 to 1.329] | 0.980 [0.912 to 1.052] | 1.200 [1.033 to 1.394] | 1.143 [0.854 to 1.528] | 1.041 [0.893 to 1.215] | 1.488 [1.162 to 1.906]
  Day 85/Early withdrawal: n=12,18,18,4,6,6: number analyzed (Participants) | 12 | 18 | 18 | 4 | 6 | 6
  Day 85/Early withdrawal: n=12,18,18,4,6,6 | 0.923 [0.821 to 1.037] | 1.032 [0.941 to 1.132] | 0.901 [0.798 to 1.017] | 0.930 [0.701 to 1.235] | 0.826 [0.727 to 0.939] | 0.946 [0.723 to 1.237]

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-SAEs and SAEs were collected up to Day 85
Description: Safety Population consisted of all randomized participants who took at least 1 dose of study intervention.
Arm/Group | Cohorts 1 and 2: Placebo SC | Cohort 1: GSK3772847 70 mg SC | Cohort 2: GSK3772847 140 mg SC | Cohorts 3 and 4: Placebo SC | Cohort 3: GSK3772847 140 mg SC in Japanese Participants | Cohort 4: GSK3772847 140 mg SC in Chinese Participants
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/18 | 0/18 | 0/4 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/18 | 0/18 | 0/4 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 3/13 | 2/18 | 3/18 | 1/4 | 2/6 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohorts 1 and 2: Placebo SC (N=13) | Cohort 1: GSK3772847 70 mg SC (N=18) | Cohort 2: GSK3772847 140 mg SC (N=18) | Cohorts 3 and 4: Placebo SC (N=4) | Cohort 3: GSK3772847 140 mg SC in Japanese Participants (N=6) | Cohort 4: GSK3772847 140 mg SC in Chinese Participants (N=6)
Headache (Nervous system disorders) | 2 | 1 | 2 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 1 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT04366349/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/49/NCT04366349/SAP_001.pdf